CLINICAL TRIAL: NCT06494241
Title: A Multi-Center Study to Evaluate the Guideline Education of Oncology Departments in Small/Middle Tier Cities and County Hospitals for Diagnosis and Treatment Improvement in Patients With Metastatic Non-small Cell Lung Cancer
Brief Title: Small/Middle Tier Cities and County Lung Cancer Quality Improvement Project (QIP) Study
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161L00048
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms
Keywords: Epidermal Growth Factor Receptor; NSCLC; Non-small cell lung cancer; Osbervational
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the molecular testing pattern in metastatic NSCLC patients after QIP; To evaluate the treatment pattern in metastatic NSCLC patients after QIP.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the implementation of standardized diagnosis and treatment practice in oncology departments of Small/Middle tier cities and County hospitals, after standardized education and implementation of lung cancer clinical practice guidelines for oncology physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, at the time of signing the informed consent.
* ECOG performance status 0-2.
* Newly pathologic diagnosed metastatic NSCLC (clinical stage IV) or recurrent metastatic NSCLC.

Exclusion Criteria:

* Be participating in other intervention clinical trials.
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
* Previous enrolment in the other QIP study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly pathologic diagnosed metastatic NSCLC (clinical stage IV) or recurrent metastatic NSCLC will be enrolled.
  Approximately 1000 patients will be enrolled from about 50 sites in China.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-11-28 (Estimated); Study Completion 2027-11-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the molecular testing pattern in metastatic NSCLC patients after QIP | Approximately 1 month after last patient in
  Molecular testing-rate for the first-line treatment: Defined as the number of participants received molecular testing for the first-line treatment divided by total participants.
To evaluate the treatment pattern in metastatic NSCLC patients after QIP | Approximately 1 month after last patient in
  TKIs first-line treatment rate: Defined as TKIs first-line treatment rate in AGA positive participants.

SECONDARY OUTCOMES:
To evaluate the clinical outcomes in metastatic NSCLC patients after QIP | Follow up approximately 24 months after last patient in
  Progression Free Survival (PFS): Defined as the time from beginning of first-line treatment to disease progression or death for any cause, whichever occurs first.
To evaluate the treatment pattern in metastatic NSCLC patients after QIP | Approximately 1 month after last patient in
  1st/2nd/3rd generation EGFR-TKIs first-line treatment rate: Defined 1st/2nd/3rd generation EGFR-TKIs first-line treatment rate in EGFR positive participants.
To evaluate the treatment pattern in metastatic NSCLC patients after QIP | Approximately 1 month after last patient in
  Immunotherapy first-line treatment rate: Defined as PD-1 or PD-L1 inhibitors first-line treatment rate in AGA negative participants.
To evaluate the clinical outcomes in metastatic NSCLC patients after QIP | Follow up approximately 24 months after last patient in
  Response rate: Defined as the percentage of participants with the disease first-line treatment response by investigator assessment as recorded in CRF.
To evaluate the clinical outcomes in metastatic NSCLC patients after QIP | Follow up approximately 24 months after last patient in
  Disease control rate: Defined as the percentage of participants with the disease first-line treatment control by investigator assessment as recorded in CRF
To evaluate the clinical outcomes in metastatic NSCLC patients after QIP | Follow up approximately 24 months after last patient in
  Duration of Response: Defined as the time from first-line treatment response to disease progression or death in participants who achieve responding by investigator assessment as recorded in CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong WU, Principal Investigator — Guangdong Provincial People's Hospital
Locations (46):
- China (46):
  - Research Site, Anning
  - Research Site, Anqing
  - Research Site, Changzhi
  - Research Site, Daqing
  - Research Site, Dazhou
  - Research Site, Dazhu
  - Research Site, Dingzhou
  - Research Site, Ganzhou
  - Research Site, Guangzhou
  - Research Site, Guang’an
  - Research Site, Hanzhong
  - Research Site, Hebi
  - Research Site, Hengyang
  - Research Site, Huaibei
  - Research Site, Jining
  - Research Site, Jinzhou
  - Research Site, Liyang
  - Research Site, Lu'an
  - Research Site, Meihekou
  - Research Site, Nanchong
  - Research Site, Nanyang
  - Research Site, Ningde
  - Research Site, Ningxiang
  - Research Site, Panjin
  - Research Site, Pingxiang
  - Research Site, Quanzhou
  - Research Site, Shengzhou
  - Research Site, Suzhou
  - Research Site, Taizhou
  - Research Site, Tancheng
  - Research Site, Tongling
  - Research Site, Wafangdian
  - Research Site, Weifang
  - Research Site, Wuzhou
  - Research Site, Xiangtan
  - Research Site, Xianning
  - Research Site, Xiantao
  - Research Site, Xixian
  - Research Site, Xuzhou
  - Research Site, Yangjiang
  - Research Site, Yangzhou
  - Research Site, Yibin
  - Research Site, Yichun
  - Research Site, Yingkou
  - Research Site, Zhangjiakou
  - Research Site, Zhuji

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/